CLINICAL TRIAL: NCT00533169
Title: A Phase I Study of ZD6474 (Zactima) Alone and in Combination With Retinoic Acid in Relapsed and Refractory Pediatric Neuroblastoma
Brief Title: ZD6474 Alone and in Combination With Retinoic Acid in Pediatric Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0807
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; ZD6474; Zactima; Isotretinoin; 13-Cis Retinoic Acid; Accutane; Pediatric Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — vandetanib; Tretinoin; Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZD6474 + Retinoic Acid (Experimental): Part A = ZD6474 Alone, Starting dose 50 mg/m^2 by mouth daily for 28 days; Part B, C = ZD6474 + Retinoic Acid 80 mg/m^2 by mouth twice daily for 2 consecutive weeks out of every four weeks (28 days).
  Interventions: Drug: ZD6474; Drug: Retinoic Acid

INTERVENTIONS:
Drug: ZD6474 — Part A = Starting dose 50 mg/m^2 by mouth daily for 28 days; Part B, C = Starting dose 50 mg/m^2 by mouth daily on days 2-28.
  Other Names: Zactima; Vandetanib
Drug: Retinoic Acid — Part B, C = 80 mg/m^2 by mouth twice daily for 2 consecutive weeks out of every four weeks (28 days).
  Other Names: Isotretinoin; Accutane; 13-cis-Retinoic Acid

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of the drug ZactimaTM (ZD6474) in patients with neuroblastoma or medulloblastoma that has gotten worse, has come back, or has not responded to the treatment.

Primary Objective:

-To determine the pharmacokinetics, safety, dose-limiting toxicities, and maximum tolerated dose of ZD6474, alone in children with medulloblastoma, and alone in combination with retinoic acid, in patients with relapsed or refractory neuroblastoma.

Secondary Objective:

-To assess progression-free survival (PFS) and objective tumor response rates in children with relapsed and refractory neuroblastoma and medulloblastoma treated with ZD6474 +/- retinoic acid in the context of a Phase I trial.

DETAILED DESCRIPTION:
The Study Drugs:

ZD6474 is a drug that slows down the function of proteins in tumor cells called protein tyrosine kinases. Tyrosine kinases normally cause tumor cells to grow. It is thought to have anti-cancer effects when given with or without other chemotherapy drugs.

Isotretinoin has been shown to help stop the growth of neuroblastoma cells. It helps cells look more normal and grow more slowly.

Study Drug Dose Level and Drug Administration:

There will be 3 parts in the study. If you have medulloblastoma, you will be assigned to Part A. If you have neuroblastoma, you will be assigned to Part A, Part B, or Part C.

In Part A, participants will receive the study drug ZD6474 alone. In the Part B portion, participants will receive ZD6474 along with isotretinoin. In Part C, an additional number of participants will be enrolled and will receive ZD6474 along with isotretinoin at the highest dose level that was found in Part B.

Part A Treatment:

Participants in Part A will take ZD6474 daily by mouth in the form of pills or liquid for 28 days. This 28-day period is called a study "cycle." In Part A, the study drug will be given at different doses. Three (3) participants will be enrolled in each dose level. New groups will continue to be enrolled at higher doses until intolerable side effects are seen. If you are assigned to Part A, the dose assigned to you will depend on the number of participants that have been enrolled before you and the side effects they may have experienced.

Part B Treatment:

Once the highest tolerable dose of ZD6474 is found, participants will then begin enrolling in Part B.

Participants in Part B will take ZD6474 daily by mouth in the form of pills or liquid on Days 2-28 of each 28-day cycle. Participants will also take isotretinoin by mouth 2 times a day every day for 2 weeks in a row, at some point during each 28-day cycle.

Part C Treatment:

In Part C, participants will follow the same schedule as in Part B.

Drug Diary (all participants):

You will be given a "diary" to record when you take the study drugs. You will need to bring the diary with you to each study visit. At each visit, you will also be asked about any side effects that you may be experiencing.

Study Visits (all participants):

During the first 2 months of the study, you will have a study visit weekly. After the first 2 months, you will have study visits at least 1 time a month.

At these visits, the following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will have a physical exam.
* Blood (about 2 teaspoons) and urine will be collected for routine tests. Before each cycle, some of the blood collection will be used for blood clotting tests. Once a month, this routine blood/urine test will include a pregnancy test for women who are able to have children.
* You will be asked about any drugs you may be taking and if you have been able to maintain a healthy diet.

Before every other cycle, the following tests and procedures will be performed:

* You may have a CT scan, MRI scan, and/or bone scan to check the status of the disease.
* You may have bone marrow aspirations and a bone marrow biopsy to check the status of the disease.
* If you have neuroblastoma, you may have an MIBG scan to check the status of the disease.
* If you have neuroblastoma, urine will be collected to test your HVA and VMA levels.

Once a week during Weeks 1, 2, 4, 9, 13, and then up to 7 days before every other cycle, you will have ECGs to make sure that your heart remains healthy.

Before each cycle, urine will be collected for routine tests and you will have an ECHO to make sure that your heart remains healthy.

Pharmacokinetic Testing:

Extra blood samples will be drawn during the study for pharmacokinetic (PK) test. PK tests are used to measure the amount of study drug in the blood. The amount of blood draw will be about 1/2 teaspoon each time.

Blood will be drawn for PK testing at the following time points:

* On Day 1 of Cycle 1, before and 6 hours after taking ZD6474
* On Days 2, 8, 15 and 22 of Cycle 1 before you take ZD6474
* On Days 1, 8 and 15 of Cycle 2 before you take ZD6474
* On Day 1 of Cycles 4, 6, and 8 before taking ZD6474

If you are 1 of the first 3 participants enrolled in the study, blood will be drawn at 2, 4, 6, and 8 or 12 and 24 hours after the very first dose during Cycle 1.

Length of Study:

You may remain on study for as long as you are benefitting. You will be taken off study early if the disease gets worse or intolerable side effects occur.

End-Of-Study Visit:

Once you are off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed. If any tests or procedure has been performed in the last month, it will not be repeated.

* Your complete medical history will be recorded.
* You will be asked about any drugs you may be taking.
* You will have a physical exam.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.
* You will have an ECHO.
* You will have an ECG.
* You may have a CT scan, MRI scan, and/or a bone scan to check the status of the disease.
* You may have bone marrow aspirations and a bone marrow biopsy to check the status of the disease.
* If you have neuroblastoma, you will have an MIBG scan to check the status of the disease.
* If you have neuroblastoma, urine will be collected to test your HVA and VMA levels.

Follow-up Visits:

You will have follow-up visits every month once you are off study. These visits will continue indefinitely. At these visits, you will have the following tests and procedures performed.

* Your complete medical history will be recorded.
* You will have a physical exam.
* Blood (about 2 teaspoons) and urine will be collected for routine tests.

This is an investigational study. ZD6474 is FDA approved for the treatment of follicular, medullary, anaplastic, and locally advanced and metastatic papillary thyroid cancer. Isotretinoin is FDA approved for acne. The use of these drugs for this disease and the use of the drugs together is investigational. Up to 66 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent from subjects or their legal guardians
2. Patients must have had histologic verification of neuroblastoma, ganglioneuroblastoma, or ganglioneuroma, and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines (Vanillylmandelic Acid (VMA) and/or Homovanillic Acid (HVA)), OR histologic verification of medulloblastoma, AND which has progressed on standard therapy, relapsed after standard therapy, or for which no standard curative therapy is known.
3. Measurable or evaluable disease presence within 4 weeks of onset of study therapy: a. measurable tumor on magnetic resonance imaging (MRI), computed tomography (CT) scan or X-ray obtained prior to study entry. Patients who appear to have residual stable tumor upon completion of frontline therapy must undergo a biopsy to document presence of viable neuroblastoma or medulloblastoma. If only active target lesion was radiated of patients with stable disease, biopsy must be done at least 4 weeks after radiation was completed and must demonstrate viable tumor, OR
4. (Con't # 3): Evaluable disease documented by bone marrow obtained prior to study entry with tumor cells seen on routine morphology (not by Neuron Specific Enolase (NSE) staining only) of aspirate and/or biopsy OR
5. (Con't # 3) (for neuroblastoma patients only) Evaluable disease documented by MIBG (metaiodobenzylguanidine) scan or bone scan obtained within 4 weeks prior to study entry with positive uptake at a minimum of one site. Patients who appear to have residual stable MIBG positive lesions upon completion of frontline therapy must undergo a biopsy to document the presence of viable neuroblastoma. If the patient has only one MIBG positive lesion and that lesion was radiated, a biopsy must be done at least 4 weeks after radiation was completed and must demonstrate viable neuroblastoma.
6. Performance status - Lansky play or karnofsky score of > / = 40
7. Age >/=2 years at time of enrollment

Exclusion Criteria:

1. Lab results: a) Absolute neutrophil count (ANC) <750/mm^3, hemoglobin <7.0 g/dL, platelets <20,000/mm^3 (hemoglobin and platelets may be supported by transfusions); b) Serum bilirubin >1.5 * institutional upper limit of normal (IULN); c) Serum creatinine >1.5 * per IULN or creatinine clearance <or equal to 70 ml/min/1.73m^2; d) Potassium, <4.0 mmol/L despite supplement; Serum calcium or ionized calcium >IULN; Magnesium out of normal range per institutional guidelines despite supplement; e) ALT > 2.5 * IULN or alkaline phosphatase (ALP) >2.5 * IULN or > 5 * IULN if judged by the investigator to be related to liver metastases
2. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
3. History of symptomatic or medically managed arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) (>/= National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation controlled on medication is not excluded.
4. Previous history of Corrected QT (QTc) prolongation as a result from other medication that required discontinuation of that medication.
5. Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age.
6. Presence of left bundle branch block
7. QTc with Bazett's correction that is unmeasurable, or >/=480 msec on screening Electrocardiography (ECG). If a patient has QTc >/=480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <480 msec in order for the patient to be eligible for the study.
8. Use of any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function
9. Clinically significant cardiac event such as myocardial infarction, TIA, or CVA within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
10. Hypertension > 95th percentile for age (either systolic or diastolic) or > 140/90 for patients >18 years of age and uncontrolled by oral medication at onset of study therapy.
11. Currently active diarrhea that may affect the ability of the patient to absorb the ZACTIMA.
12. Women who are currently pregnant or breastfeeding.
13. Receipt of any investigational agents within 14 days prior to commencing study treatment, or prior receipt of ZACTIMA at any time
14. Last dose of prior chemotherapy discontinued less than 2 weeks before the start of study therapy.
15. Last radiation therapy within the last 4 weeks before the start of study therapy, except palliative radiotherapy to non-index lesions
16. Any unresolved non-hematologic toxicity greater than CTC grade 1 from previous anti-cancer therapy, except for platinum-induced hearing loss.
17. Any evidence of active graft versus host disease after stem cell transplant.
18. Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 day cycles, first 2 cycles used to determine dose-limiting toxicity
  MTD is highest dose level in which 6 participants have been treated with at most 2 experiencing dose limiting toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Peter E. Zage, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org